CLINICAL TRIAL: NCT01350102
Title: The Relationship of Hemoglobin A1c and Diabetic Wound Healing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study closed due to recruitment problems
Sponsor: Susan Hassenbein (Other)
Responsible Party: Sponsor-Investigator, Susan Hassenbein, Clinical Research Associate, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-35832
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Diabetes, Type 1; Diabetes, Type 2; Foot Ulcer, Diabetic
Keywords: Adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Foot | interventions — Bacitracin; oak bark extract; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bacitracin wound care dressing alone (Active Comparator): Bacitracin wound care dressing alone
  Interventions: Drug: Bacitracin
- Bacitracin with Vit C (Active Comparator): Bacitracin wound care dressing with Vitamin C supplementation
  Interventions: Drug: Bacitracin; Dietary Supplement: Vitamin C
- AmeriGel® wound care dressing alone (Active Comparator): AmeriGel® wound care dressing alone
  Interventions: Drug: AmeriGel®
- AmeriGel® with Vit C (Active Comparator): AmeriGel® wound care dressing with Vitamin C supplementation
  Interventions: Drug: AmeriGel®; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Bacitracin — Participants will be treated with Bacitracin to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Other Names: Baciguent
  Arms: Bacitracin with Vit C; Bacitracin wound care dressing alone
Drug: AmeriGel® — Participants will be treated with AmeriGel® to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Other Names: Oakin®-based hydrogel; hydrogel containing Oakin®; Oak extract
  Arms: AmeriGel® with Vit C; AmeriGel® wound care dressing alone
Dietary Supplement: Vitamin C — Participants will be treated with Vitamin C supplements 1000 mg daily until 100% wound healing, which may take up to 6 months to achieve
  Other Names: ascorbic acid
  Arms: AmeriGel® with Vit C; Bacitracin with Vit C

SUMMARY:
The purpose of this study is to investigate the relationship of hemoglobin A1c in diabetic wound healing. Additionally, a comparison of two wound dressings, AmeriGel® (Amerx Health Care Corp., Clearwater, FL) and Bacitracin, with and without vitamin C supplementation, will be done to evaluate impact on time to wound closure.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study evaluating the relationship of hemoglobin A1c in diabetic wound healing. Length of time for wound closure will be compared using four treatment options.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diabetic (Type I and Type II)
* Ulceration of the foot at least one centimeter in width/length
* Ulceration at least 0.2 centimeters in depth

Exclusion Criteria:

* Ulceration width/length > 7.5 centimeters
* Wound depth > 1.25 centimeters
* Purulent, excessive drainage and/or other signs of infection (i.e. erythema, edema, warmth)
* Inability to provide informed consent
* Inability to swallow pills (vitamin C supplement)
* Patients with concurrent renal problems
* Patients with medication contraindications to Vitamin C and/or topical wound dressings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nell V. Blake, DPM, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markuson M, Hanson D, Anderson J, Langemo D, Hunter S, Thompson P, Paulson R, Rustvang D. The relationship between hemoglobin A(1c) values and healing time for lower extremity ulcers in individuals with diabetes. Adv Skin Wound Care. 2009 Aug;22(8):365-72. doi: 10.1097/01.ASW.0000358639.45784.cd. PMID 19638800
- [Background] Jensen JL, Seeley J, Gillin B. Diabetic foot ulcerations. A controlled, randomized comparison of two moist wound healing protocols: Carrasyn Hydrogel Wound dressing and wet-to-moist saline gauze. Adv Wound Care. 1998 Nov-Dec;11(7 Suppl):1-4. No abstract available. PMID 10326334
- [Background] Storm DR. Mechanism of bacitracin action: a specific lipid-peptide interaction. Ann N Y Acad Sci. 1974 May 10;235(0):387-98. doi: 10.1111/j.1749-6632.1974.tb43278.x. No abstract available. PMID 4368896
- [Background] Falabella A, Falanga V. Uncommon causes of ulcers. Clin Plast Surg. 1998 Jul;25(3):467-79. PMID 9696906
- [Background] Lazarus GS, Cooper DM, Knighton DR, Margolis DJ, Pecoraro RE, Rodeheaver G, Robson MC. Definitions and guidelines for assessment of wounds and evaluation of healing. Arch Dermatol. 1994 Apr;130(4):489-93. PMID 8166487
- [Background] Maklebust JA, Margolis D. The goodness of measurement. Adv Wound Care. 1996 May-Jun;9(3):6. No abstract available. PMID 8716267
- [Background] van Rijuswijl L. Wound assessment and documentation. In: Krasner LD, Rodeheaver GT, Sibbald RG (eds). Chronic Wound Care: A Clinical Source Book for Healthcare Professionals, 3rd ed. Wayne Pa: HMP Communications: 2001;101-115.
- [Background] Keast DH, Bowering CK, Evans AW, Mackean GL, Burrows C, D'Souza L. MEASURE: A proposed assessment framework for developing best practice recommendations for wound assessment. Wound Repair Regen. 2004 May-Jun;12(3 Suppl):S1-17. doi: 10.1111/j.1067-1927.2004.0123S1.x. PMID 15230830
- [Background] Haslik W, Kamolz LP, Andel H, Winter W, Meissl G, Frey M. The influence of dressings and ointments on the qualitative and quantitative evaluation of burn wounds by ICG video-angiography: an experimental setup. Burns. 2004 May;30(3):232-5. doi: 10.1016/j.burns.2003.10.016. PMID 15082349
- [Background] Droog EJ, Steenbergen W, Sjoberg F. Measurement of depth of burns by laser Doppler perfusion imaging. Burns. 2001 Sep;27(6):561-8. doi: 10.1016/s0305-4179(01)00021-3. PMID 11525849
- [Background] Duckworth WC, Fawcett J, Reddy S, Page JC. Insulin-degrading activity in wound fluid. J Clin Endocrinol Metab. 2004 Feb;89(2):847-51. doi: 10.1210/jc.2003-031371. PMID 14764804
- [Background] Zimny S, Schatz H, Pfohl M. Determinants and estimation of healing times in diabetic foot ulcers. J Diabetes Complications. 2002 Sep-Oct;16(5):327-32. doi: 10.1016/s1056-8727(01)00217-3. PMID 12200075
- [Background] Rubinstein A, Pierce CE Jr. Rapid healing of diabetic foot ulcers with meticulous blood glucose control. Acta Diabetol Lat. 1988 Jan-Mar;25(1):25-32. doi: 10.1007/BF02581242. PMID 3043987
- [Background] Yue DK, McLennan S, Marsh M, Mai YW, Spaliviero J, Delbridge L, Reeve T, Turtle JR. Effects of experimental diabetes, uremia, and malnutrition on wound healing. Diabetes. 1987 Mar;36(3):295-9. doi: 10.2337/diab.36.3.295. PMID 3803737
- [Background] Vitamin C and the common cold. Med Lett Drugs Ther. 1970 Dec 25;12(26):105-6. No abstract available. PMID 4936077
- [Background] Howe GR, Hirohata T, Hislop TG, Iscovich JM, Yuan JM, Katsouyanni K, Lubin F, Marubini E, Modan B, Rohan T, et al. Dietary factors and risk of breast cancer: combined analysis of 12 case-control studies. J Natl Cancer Inst. 1990 Apr 4;82(7):561-9. doi: 10.1093/jnci/82.7.561. PMID 2156081
- [Background] Wassertheil-Smoller S, Romney SL, Wylie-Rosett J, Slagle S, Miller G, Lucido D, Duttagupta C, Palan PR. Dietary vitamin C and uterine cervical dysplasia. Am J Epidemiol. 1981 Nov;114(5):714-24. doi: 10.1093/oxfordjournals.aje.a113243. PMID 7304600
- [Background] Snyder RJ, Kirsner RS, Warriner RA 3rd, Lavery LA, Hanft JR, Sheehan P. Consensus recommendations on advancing the standard of care for treating neuropathic foot ulcers in patients with diabetes. Ostomy Wound Manage. 2010 Apr;56(4 Suppl):S1-24. PMID 20424290
- [Background] Pollack SV. Wound healing: a review. III. Nutritional factors affecting wound healing. J Dermatol Surg Oncol. 1979 Aug;5(8):615-9. doi: 10.1111/j.1524-4725.1979.tb00733.x. PMID 479447
- [Background] van Anholt RD, Sobotka L, Meijer EP, Heyman H, Groen HW, Topinkova E, van Leen M, Schols JM. Specific nutritional support accelerates pressure ulcer healing and reduces wound care intensity in non-malnourished patients. Nutrition. 2010 Sep;26(9):867-72. doi: 10.1016/j.nut.2010.05.009. Epub 2010 Jul 3. PMID 20598855
- [Background] Smith RG. Validation of Wagner's classification: a literature review. Ostomy Wound Manage. 2003 Jan;49(1):54-62. PMID 12532034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two subjects were screened and enrolled at the clinic site on 2/24/2012 and 1/14/2013.
Groups:
- Bacitracin Wound Care Dressing Alone: Bacitracin wound care dressing alone
  Bacitracin: Participants will be treated with Bacitracin to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Hemoglobin A1c: Hemoglobin A1c levels will be performed and reviewed every three months to assess its relationship to wound healing
- Bacitracin With Vit C: Bacitracin wound care dressing with Vitamin C supplementation
  Bacitracin: Participants will be treated with Bacitracin to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Hemoglobin A1c: Hemoglobin A1c levels will be performed and reviewed every three months to assess its relationship to wound healing
  Vitamin C: Participants will be treated with Vitamin C supplements 1000 mg daily until 100% wound healing, which may take up to 6 months to achieve
- AmeriGel® Wound Care Dressing Alone: AmeriGel® wound care dressing alone
  AmeriGel®: Participants will be treated with AmeriGel® to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Hemoglobin A1c: Hemoglobin A1c levels will be performed and reviewed every three months to assess its relationship to wound healing
- AmeriGel® With Vit C: AmeriGel® wound care dressing with Vitamin C supplementation
  AmeriGel®: Participants will be treated with AmeriGel® to their wound until 100% wound healing, which may take up to 6 months to achieve.
  Hemoglobin A1c: Hemoglobin A1c levels will be performed and reviewed every three months to assess its relationship to wound healing
  Vitamin C: Participants will be treated with Vitamin C supplements 1000 mg daily until 100% wound healing, which may take up to 6 months to achieve
Period: Overall Study
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C
Started | 0 | 1 | 1 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C | Total
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Hgb A1c Level
Description: Hgb A1c measures the average blood glucose over three months (% of hemoglobin). All subjects will be asked to get their hemoglobin A1c level at the beginning of the study and every three months for as long as they participate in the study.
Time Frame: Patients are assessed every 3 months from enrollment through end of study participation, which may be 6 months
Population: Enrollment and 3-month visit A1c levels were obtained for the subject in the Bacitracin with Vit C arm. Enrollment A1c level was obtained for the AmeriGel would care dressing alone.
  However, this subject withdrew from the study before 3-month A1c level was obtained.
Measure: Number; unit: percentage of hemoglobin
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C
Number analyzed (Participants) | 0 | 1 | 1 | 0
percentage of hemoglobin
  Enrollment A1c |  | 5.2 | 12.1 |
  3 Month A1c |  | 6.1 | NA — A1c not taken - patient withdrawn from study prior to 3 months |

2. Secondary Outcome: Length of Time for Wound Closure
Description: Length of time for wound closure will be measured in days
Time Frame: Patients are assessed every other week (bi-weekly) until 100% wound healing is achieved, which may take up to 6 months
Population: Only the subject in the Bacitracin with Vit C arm achieved would healing. The subject in the AmeriGel would care dressing alone arm was withdrawn due to lack of healing and infection.
Measure: Number; unit: Days
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C
Number analyzed (Participants) | 0 | 1 | 0 | 0
Days |  | 141 |  |

3. Secondary Outcome: Wound Area Measurements
Description: Wound area measurements in length, width, and depth throughout the course of the study(measured in cm).
Time Frame: Patients are assessed every other week (bi-weekly) until 100% wound healing is achieved, which may take up to 6 months
Population: The subject enrolled in Bacitracin with Vit C arm had measurements of the wound (width, depth, length) recorded beginning at week 0 through week 20. The subject enrolled in the AmeriGel wound care dressing alone had measurements recorded of the wound (width, depth, length) beginning at week 0 through week 2 before withdrawing from the study.
Measure: Number; unit: cm
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C
Number analyzed (Participants) | 0 | 1 | 1 | 0
cm
  Week 0 Width of Wound |  | 0.9 | 0.3 |
  Week 0 Depth of Wound |  | 0.2 | 0.2 |
  Week 0 Length of Wound |  | 1.0 | 2 |
  Week 2 Width of Wound |  | 0.4 | 0.5 |
  Week 2 Depth of Wound |  | 0.1 | 0.2 |
  Week 2 Length of Wound |  | 0.5 | 0.5 |
  Week 4 Width of Wound |  | 0.4 | NA — Withdrawn from study |
  Week 4 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 4 Length of Wound |  | 0.5 | NA — Withdrawn from study |
  Week 6 Width of Wound |  | 0.2 | NA — Withdrawn from study |
  Week 6 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 6 Length of Wound |  | 0.2 | NA — Withdrawn from study |
  Week 8 Width of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 8 Depth of Wound |  | 0.3 | NA — Withdrawn from study |
  Week 8 Length of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 10 Width of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 10 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 10 Length of Wound |  | 0.2 | NA — Withdrawn from study |
  Week 12 Width of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 12 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 12 Length of Wound |  | 0.3 | NA — Withdrawn from study |
  Week 14 Width of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 14 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 14 Length of Wound |  | 0.3 | NA — Withdrawn from study |
  Week 16 Width of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 16 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 16 Length of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 18 Width of Wound |  | 0.3 | NA — Withdrawn from study |
  Week 18 Depth of Wound |  | 0.1 | NA — Withdrawn from study |
  Week 18 Length of Wound |  | 0.3 | NA — Withdrawn from study |
  Week 20 Width of Wound |  | 0.0 | NA — Withdrawn from study |
  Week 20 Depth of Wound |  | 0.0 | NA — Withdrawn from study |
  Week 20 Length of Wound |  | 0.0 | NA — Withdrawn from study |

ADVERSE EVENTS:
Time Frame: enrollment through 20 weeks
Arm/Group | Bacitracin Wound Care Dressing Alone | Bacitracin With Vit C | AmeriGel® Wound Care Dressing Alone | AmeriGel® With Vit C
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bacitracin Wound Care Dressing Alone (N=0) | Bacitracin With Vit C (N=1) | AmeriGel® Wound Care Dressing Alone (N=1) | AmeriGel® With Vit C (N=0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Wound infection at 2 weeks; patient withdrawn from study and provided standard of care treatment to include antibiotics.

LIMITATIONS AND CAVEATS:
Study terminated due to recruitment issues - only two subjects enrolled in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes